CLINICAL TRIAL: NCT04330430
Title: Neo-adjuvant T-VEC + Nivolumab Combination Therapy for Resectable Early Metastatic (stage IIIB/C/D-IV M1a) Melanoma with Injectable Disease
Acronym: NIVEC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N19TVN
Record Dates: First submitted 2020-02-13; First posted 2020-04-01 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Melanoma Stage III; Melanoma Stage IV
Keywords: Melanoma; Neo-adjuvant; T-VEC; Nivolumab
MeSH Terms: conditions — Melanoma | interventions — talimogene laherparepvec; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- T-VEC + Nivolumab (Experimental): Patients will receive pre-surgically 4 courses T-VEC (up to 4ml; first dose 10^6 PFU per mL, subsequent doses at 10^8 PFU per mL). Patients will also receive a flatdose of 240mg Nivolumab every 2 weeks after the first T-VEC injections (starting at 2nd T-VEC course at week 3, followed by the next doses at week 5 and 7).
  Interventions: Drug: T-VEC

INTERVENTIONS:
Drug: T-VEC — The treatment schedule is based on 4 courses of intralesional T-VEC and 3 courses of intraveneous Nivolumab. T-VEC first, in order to achieve the best synergistic effect with influx of CD8+ T-cells prior to the first Nivolumab dose. T-VEC monotherapy with the dose 10^8 PFU/mL is given every 2 weeks after 3 weeks of the first T-VEC dose (with the first dose of T-VEC 10^6 PFU/mL to allow for seroconversion), and Nivolumab will be given every 2 weeks.
  Other Names: Nivolumab

SUMMARY:
Currently, standard treatment options available for Stage III melanoma include locoregional management (i.e. surgery) or systemic treatment (adjuvant to surgery or primarily in the case of unresectable disease).

Adjuvant treatment options have shown major improvements in overall survival (OS) and relapse free survival (RFS) in resected stage III or IV melanoma.

In daily practice, T-VEC monotherapy is used for unresectable Stage IIIB-IVM1a (injectable) disease, whereas Nivolumab is used for stage IV melanoma (among other systemic therapies).

The next major developments are in neo-adjuvant treatment options for resectable stage III disease, where 3 small studies reported high response rates with systemic immunotherapy.

This study evaluates the combination treatment of T-VEC + Nivolumab in the neo-adjuvant setting. The concept is that T-VEC can turn an immune desolate "cold" tumor into an immunogenic "hot" tumor. The hypothesis is that this will upregulate the expression of PD-L1 and make it more susceptible for treatment with an anti-PD-1 agent. The investigators believe neo-adjuvant Nivolumab + T-VEC will thus change the tumor microenvironment in patients with stage IIIB/C/D/IVM1a (AJCC 8) melanoma with resectable cutaneous or subcutaneous satellite or in-transit metastases (ITM) and/or tumor positive lymph nodes. With this trial the investigators aim to determine safety and feasibility of combination neo-adjuvant Nivolumab + T-VEC in patients with stage III melanoma with resectable ITM and/or tumor positive lymph nodes. The treatment schedule is based on 4 courses of intralesional T-VEC and 3 courses of intravenous Nivolumab. T-VEC first, in order to achieve the best synergistic effect with influx of CD8+ T cells prior to the first Nivolumab dose. T-VEC monotherapy with the dose 108 PFU/mL is given every 2 weeks (± 3) days after 3 weeks of the first T-VEC dose (with the first dose of T-VEC 106 PFU/mL to allow for seroconversion) , and Nivolumab can be given either every 2 weeks or every 4 weeks. Therefore we suggest the same dosing schedule for T-VEC and Nivolumab every 2 weeks for the purpose of this trial.

ELIGIBILITY:
Inclusion Criteria:

* Adults at least 18 years of age
* WHO performance score of 0 or 1
* Cytologically or histologically confirmed diagnosis of stage IIIB/C/D/IVM1a (AJCC 8th edition) melanoma, eligible for surgical resection.
* Subjects must have measurable disease according to RECIST 1.1 and must be a candidate for intralesional therapy with at least one injectable cutaneous, subcutane-ous or nodal melanoma lesion (≥ 10 mm in longest diameter) or with multiple injectable lesions that in aggregate have a longest diameter of ≥ 10 mm.
* Prior isolated limb perfusion (ILP) is allowed (≥ 12 weeks prior to enrolment)
* Screening laboratory values must meet the following criteria:
* WBC ≥ 2.0x10^9/L, Neutrophils ≥1.5x10^9/L, Platelets ≥100 x10^9/L, Hemoglobin ≥5.5 mmol/L, Creatinine ≤1.5x ULN, AST ≤ 1.5 x ULN, ALT ≤ 1.5 x ULN, Bilirubin ≤1.5 X ULN
* LDH < 2 x ULN
* Women of childbearing potential (WOCBP) must use highly effective method(s) of contraception (see paragraph 5.2) during T-VEC and nivolumab treatment and for a period of 5 months after the last dose of nivolumab.
* Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to enrollment and within 24 hours prior to the start of Nivolumab
* Men receiving nivolumab and who are sexually active with WOCBP should use contraception during treatment and for a period of 7 months after the last dose of nivolumab
* Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year.
* Women who are not of childbearing potential (i.e., who are postmenopausal), or surgically sterile as well as azoospermic men do not require contraception
* Patient is capable of understanding and complying with the protocol requirements and has signed the Informed Consent document.
* Inhaled or topical steroids, and adrenal replacement steroid < 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease
* International normalization ratio (INR) or prothrombin time (PT) ≤1.5 x ULN, unless the subject is receiving anticoagulant therapy, in which case PT and partial thrombo-plastin time (PTT)/ activated PTT (aPTT) must be within therapeutic range of intended use of anticoagulants.

Exclusion Criteria:

* Liver, Bone, Lung, Brain or other Visceral Metastases.
* No measurable lesion according to RECIST 1.1
* Prior radiotherapy for melanoma
* Prior systemic cancer therapies, including, but not limited to anti-CTLA-4, anti-PD-1, anti-PD-L1
* No other malignancies, except adequately treated and a cancer-related life-expectancy of more than 5 years.
* Patients will be excluded if they test positive for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody), indicating acute or chronic infection
* Patients will be excluded if they have known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* History or evidence of active autoimmune disease that requires high dose systemic treatment (ie, with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic cortico-steroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Evidence of clinically significant immunosuppression such as the following:
* Primary immunodeficiency state such as Severe Combined Immunodeficiency Dis-ease.
* Concurrent opportunistic infection.
* Receiving systemic immunosuppressive therapy (> 2 weeks) including oral steroid doses > 10 mg/day of prednisone or equivalent within 7 days prior to enrollment
* Active herpetic skin lesions or prior complications of HSV-1 infection (e.g., herpetic keratitis or encephalitis).
* Requirement of intermittent or chronic systemic (intravenous or oral) treatment with an antiherpetic drug (e.g., acyclovir), other than intermittent topical use.
* Previous treatment with talimogene laherparepvec or any other oncolytic virus.
* Received live vaccine within 30 days prior to enrollment.
* Subject has known sensitivity to talimogene laherparepvec or nivolumab or any of its components to be administered during dosing.
* Female subject of childbearing potential who is unwilling to use highly effective meth-od(s) of effective contraception during study treatment and through 5 months after the last dose of study medication (per protocol through 3 months after the last dose of talimogene laherparepvec and through 5 months after the last dose of nivolumab).
* Sexually active subjects and their partners unwilling to use male or female latex condom to avoid potential viral transmission during sexual contact while on treatment and within 30 days after treatment with talimogene laherparepvec.
* Subjects who are unwilling to minimize exposure with his/her blood or other body flu-ids to individuals who are at higher risks for HSV-1 induced complications such as immunosuppressed individuals, individuals known to have HIV infection, pregnant women, or infants under the age of 3 months, during talimogene laherparepvec treatment and through 30 days after the last dose of talimogene laherparepvec.
* No Allergies and Adverse Drug Reaction
* History of allergy to study drug components
* History of severe hypersensitivity reaction to any monoclonal antibody
* No underlying medical conditions that, in the Investigator's opinion, will make the ad-ministration of study drug hazardous or obscure the interpretation of toxicity determination or adverse events;
* No use of other investigational drugs before study drug administration 30 days and 5 half-times before study inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2023-04-09 (Actual); Study Completion 2025-01-29 (Actual)

PRIMARY OUTCOMES:
Pathologic response | 12 weeks
  Pathologic response according to central revision by pathology of NKI (complete response, near complete response (<10% vital tumor remaining)

SECONDARY OUTCOMES:
Rate of delay of surgery > 14 days | 9 weeks
Rate of failure to perform surgery defined as no surgery at all (due to progressive disease or adverse events) | 9 weeks
Relapse free survival (RFS) | Up to 2 years after treatment
  Relapse free survival as defined from date of surgery until date of first relapse (regardless of site)
Safety of neo-adjuvant combination of T-VEC and nivolumab according to CTCAE v5.0 | 12 weeks
Acquiring tumor tissue | Up to 2 years after treatment
  The objective is to acquire tumor tissue for prognostic biomarker research, for example CD8
Acquiring tumor tissue | Up to 2 years after treatment
  The objective is to acquire tumor tissue for prognostic biomarker research, for example IFN-γ
Acquiring tumor tissue | Up to 2 years after treatment
  The objective is to acquire tumor tissue for prognostic biomarker research, for example PD-L1
Acquiring tumor tissue | Up to 2 years after treatment
  The objective is to acquire tumor tissue for exploration of expansion of tumor-resident T cells in the tumor

CONTACTS AND LOCATIONS:
Overall Officials: John Haanen, Prof., Principal Investigator — Medical oncologist/researcher
Locations (1):
- Antoni van Leeuwenhoek ziekenhuis, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rohaan MW, Stahlie EHA, Franke V, Zijlker LP, Wilgenhof S, van der Noort V, van Akkooi ACJ, Haanen JBAG. Neoadjuvant nivolumab + T-VEC combination therapy for resectable early stage or metastatic (IIIB-IVM1a) melanoma with injectable disease: study protocol of the NIVEC trial. BMC Cancer. 2022 Aug 4;22(1):851. doi: 10.1186/s12885-022-09896-4. PMID 35927710